CLINICAL TRIAL: NCT03728907
Title: A Comparison of User-adjusted and Audiologist-adjusted Hearing Amplification
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We did not receive the equipment from our subcontractor in a time frame that would allow us to complete the study.
Sponsor: San Diego State University (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Carol L Mackersie, Professor, San Diego State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2183099
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Hearing Loss
Keywords: hearing aid; self-fitting
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: Repeated-measures crossover design
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcomes assessors and participants will not be aware of which hearing setting (audiologist adjusted vs. self-adjusted) they are wearing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Audiologist-adjusted first (Active Comparator): This arm will complete the field trial with the audiologist-adjusted fitting first, followed by the user-adjustment fitting.
  Interventions: Device: Hearing aid fitting technique- audiologist or user-adjusted
- User-adjusted first (Experimental): This arm will complete the trial with the user-adjusted fitting first followed by the audiologist-adjusted fitting.
  Interventions: Device: Hearing aid fitting technique- audiologist or user-adjusted

INTERVENTIONS:
Device: Hearing aid fitting technique- audiologist or user-adjusted — See information under 'arm' description

SUMMARY:
Fifty adults with mild to moderately severe sensorineural hearing loss will be fit with hearing amplification using two adjustment techniques. For the "audiologist fitting" technique, a licensed audiologist will adjust the hearing device using the standard of care procedures which include adjustment and verification of output to match prescribed targets (NAL-NL2) and subsequent fine tuning to optimize adjustments based on participant feedback. The second technique is "user-adjustment" of the device consisting of adjustment to overall level, high-frequency boost, and low-frequency cut by the participant while listening to speech. A cross-over design will be used in which half the participants are initially fit using the audiologist technique and the other half are initially fit using the user self-adjustment technique. Following a seven-day field trial, participants will return to the lab and the aids will be reset use the other technique. Participants will be blinded to the condition. During each seven-day field trial, users will have access to a volume control, Following the end of the two trials, participants will return to the lab for outcome assessment.

ELIGIBILITY:
Inclusion Criteria:

* bilateral hearing loss with a minimum of 40 dB HL thresholds at 2000 Hz
* English speaking

Exclusion Criteria:

* Score less than 21 on the MoCa (Montreal Cognitive Assessment)
* Evidence of conductive or retrocochlear pathology

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Real-ear aided output | two weeks
  aided output (in dB SPL) measured across frequencies in the ears of the participants

SECONDARY OUTCOMES:
Device Oriented Scale of Improvement (DOSO) | two weeks
  Questionnaire (25 items) to assess benefit from hearing aids on a 7 pt scale; a larger number is associated with better outcome
Computerized Assisted Speech Perception Assessment (CASPA) | two weeks
  Speech recognition test; phoneme recognition score as percentage correct

IPD SHARING:
Plan to Share IPD: No